CLINICAL TRIAL: NCT05205824
Title: Validation IMU and EMG Algorithms in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roessingh Research and Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-8218
Record Dates: First submitted 2021-12-21; First posted 2022-01-25 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Algorithm validation (Other): all subjects will be measured with inertial measurement units while performing tasks like walking, standing and sitting.
  Interventions: Other: algorithm validation

INTERVENTIONS:
Other: algorithm validation — stroke subjects are measured to validate algorithms previously developed after including healthy subjects

SUMMARY:
The objective is to validate the algorithms for movement analysis that were developed previously in healthy participants, in a small study with stroke patients. Stroke subjects will be measured while performing tasks like walking, sitting and standing while wearing light-weight inertial measurements units (IMUs) incorporating 3D accelerometers, 3D gyroscopes and surface electromyography. During the measurements subjects will be recorded on video that serves as ground truth when validating the implemented algorithms for movement analysis. A face blurring program will be used for all video footage.

DETAILED DESCRIPTION:
Subjects will perform the following tasks: 30 sec stationary sitting/standing/lying; 10m walk test; L-test; 8-figure walking test; daily life task; stepping over small obstacles; walk in the corridor. During the measurments IMU will be placed at: sternum; sacrum; bilateral wrists; bilateral shanks; bilateral upper legs; both feet. Surface EMG of bilateral rectus femoris; vastus lateralis; medial gastrocnemius and soleus will be measured.

ELIGIBILITY:
Inclusion Criteria:

* min 18 yrs of age; history of previous stroke; unilateral affected;able to walk without supervision (FAC-score min 4);able to perform activities of daily living without assistance (self-reported); written informed consent.

Exclusion Criteria:

* subjects with neurological or motor disorders that could interfere with the measurements (other than stroke) or severe deficits in communication, memory and understanding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Inertial measurement unit data | 1-2 hours
  Activity data of the sensors attached to various body parts

SECONDARY OUTCOMES:
surface EMG-data | 1-2 hours
  rectus femoris/vastus lateralis/gastrocnemius/soleus data

OTHER OUTCOMES:
anonymized video data | 1-2 hours
  Video data of the measurements performed
Age | at inclusion
  Age (in years)
Height | at inclusion
  Height (in cm)
Leg length | at inclusion
  Leg length (in cm)
Time since stroke | at inclusion
  time since stroke (in years)
Type of stroke | at inclusion
  type of stroke (ischemic or hemorrhagic)
Body side | at inclusion
  Affected and dominant body side (left or right)
FAC-score | at inclusion
  Functional Ambulation Categories score (0-5 points) to assess independence of walking
Motricity Index | at inclusion
  Motricity index lower limb (0-33 points)

CONTACTS AND LOCATIONS:
Overall Officials: C Nikamp, PhD, Principal Investigator — Roessingh Research and Development
Locations (1):
- Roessingh Research and Development, Enschede, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
not decided within the consortium yet